CLINICAL TRIAL: NCT06066229
Title: The Patient at the Center of Lung Transplantation Research - Identification of Patient Important Outcomes in Lung Transplantation
Brief Title: Identification of Patient Important Outcomes in Lung Transplantation
Acronym: PACRET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 220838
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Lung Transplant
Keywords: Lung transplantation; Patient-Important Outcomes; Patient-Reported Outcomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lung transplant patients: Adult lung transplant patients followed at Hôpital Bichat (Paris) or Hôpital Foch (Suresnes)
  Interventions: Other: Questionnaire- Delphi method
- Relatives of lung transplant patients: Close relatives of lung transplant patients (spouse; partner; first-degree parent) followed at Bichat Hospital (Paris) or Foch Hospital (Suresnes).
  Interventions: Other: Questionnaire- Delphi method
- Physicians from lung transplant: Physicians from lung transplant centers in France, or French-speaking experts identified in the professional network of investigators
  Interventions: Other: Questionnaire- Delphi method
- Paramedical staff: Nurses, psychologists, physiotherapists, etc.) from the same French center or French-speaking centers whose primary focus is on caring for lung transplant patients
  Interventions: Other: Questionnaire- Delphi method

INTERVENTIONS:
Other: Questionnaire- Delphi method — Identify important evaluation criteria for lung transplant patients by rating each criterion

SUMMARY:
Lung transplantation (LT) is the treatment for end-stage respiratory failure, for severe cases after thorough clinical and paraclinical evaluation. Patients often face a lengthy journey before being placed on the transplant list, and post-transplant care can seem to be demanding.

Patient-Important Outcomes (PIO), have emerged across various medical fields, aiming to prioritize the patient's perspective in medical research. This approach seeks to align clinical outcomes with those important to patients, such as pain, mobility, autonomy, and quality of life.

The focus on patient-centered research is crucial not only in medical care but also in clinical research. While several medical fields have embraced this approach, including diabetology, rheumatology, urology, and more, the field of lung transplantation has yet to fully explore the importance of PIO.

LT addresses diverse underlying conditions (e.g., cystic fibrosis, pulmonary fibrosis, emphysema, pulmonary hypertension), impacting potentially different patient populations. However, the transplantation process standardizes certain aspects, such as follow-up obligations, treatments, side effects, and complications, which can affect patient quality of life.

A systematic literature review of LT studies published in 2019 found that only 11 out of 51 studies evaluated PIOs beyond mortality. This highlights the need to assess interventions in this field based on criteria important to patients.

Besides the impact on the patient, the influence on their close family members and caregivers is significant. The transition from severe respiratory disease to near-normal respiratory function can lead to a reevaluation of the caregiver's role and responsibilities.

Currently, researchers and clinicians in transplantation focus more on Patient-Reported Outcomes (PRO) than on outcomes important to patients. To bridge this gap, this study aims to identify PIOs from the perspectives of clinicians, transplant recipients, and their families.

The Delphi method is chosen to gather anonymous expert opinions and reach a consensus on defining PIOs in the context of lung transplantation.

Ultimately, this research aims to create a "core outcome set" necessary for LT research, incorporating dimensions beyond mortality, which is the traditional focus in assessing transplant outcomes.

DETAILED DESCRIPTION:
Lung transplantation (LT) is an exceptional treatment for severe patients. It is a lengthy process, and its outcomes may seem burdensome. LT is the subject of thriving research: a search on ClinicalTrials with the terms 'Lung Transplant' retrieves 85 ongoing studies. Outcome measures (OM) are used to assess the impact of an intervention during a prognostic study. They must be carefully chosen, relevant, reproducible, and validated. It is challenging for researchers to find a balance between these OM, which should be objective, reliable, easily evaluable, and OM that are important to the patient (patient-important outcomes - PIO) and integrate into their daily lives. The emergence of PIO has occurred in many fields (Dinglas Thorax 2018, Partridge Lancet 2004). They 'reflect what the patient feels, their functional state, or under what conditions they survive' (Wittes, Stat Med 1989) and cover various domains (pain, mobility, autonomy, quality of life, etc.). The role of PIO in LT has never been evaluated. We conducted a systematic review aiming to describe the role of PIO in LT research, published in 2019 (Weisenburger et al., Respir Med Res 2022). At least one PIO was used in 26 out of the 51 included studies, with only 11 evaluating a PIO other than mortality. Some transplant physicians are well aware of this gap (Lamas, NEJM 2018). Placing the patient's concerns at the center is considered an essential objective in patient care and clinical research, including in LT. PIO could encompass mortality and patient-reported OM (PROMS), but there could also be OM that we, clinicians and researchers, have not considered, which could be crucial for patients. Gathering the opinions of lung transplant patients, their families, and healthcare providers (physicians and paramedics) involved in LT will help define a set of PIO in LT. This work proposes an original approach to identify PIO in LT in order to define a 'core outcome set,' a recommended set of outcome measures to be used. The development of a 'core outcome set' incorporating PIO can only be achieved through the participation of patients (Needham, AJRCCM 2017) in collaboration with clinicians and researchers. A Delphi-like methodology allows for the establishment of such criteria. Involving patients and their families places their concerns at the center of research that affects them. The two participating LT centers complement each other in terms of patient recruitment (preferentially patients with chronic obstructive bronchopneumopathy or fibrosing pneumopathies at Bichat Hospital; preferentially younger patients with cystic fibrosis at Foch Hospital). The development of a 'core outcome set' will guide the LT research community towards the selection of relevant OM for patients and healthcare providers. Such work would also involve patients and their families, which is important in the field of LT research. Our results could be used to provide recommendations for future LT research and help standardize prognostic evaluation measures. The methods for assessing the performance of LT centers could be reviewed and not solely rely on the isolated measurement of mortality." Practical implementation: A Delphi survey will be conducted. This method aims to gather anonymous opinions from one or more groups of experts in order to reach a consensus on subjects with uncertain definitions (Linstone et al. 2002; Fink et al. Am J Public Health 1984).

This methodology has been used, among others, to identify important evaluation domains for survivors of acute respiratory distress syndrome and their families (Dinglas, Thorax 2018).

Formation of four panels:

* Patients followed in one of the two participating centers (Bichat Hospital, Paris; Foch Hospital, Suresnes).
* Relatives (spouses, partners, or, if not available, first-degree relatives) of patients in one of the participating centers.
* Clinician doctors and researchers from LT centers, belonging to the lung transplantation group of the French Language Pneumology Society or the francophone network of investigators.
* Paramedical caregivers (nurses, advanced practice nurses, transplantation coordination nurses, psychologists, physiotherapists, etc.) working in one of the French or identified French-speaking centers.

ELIGIBILITY:
Inclusion Criteria:

Lung transplant patients followed at Bichat Hospital (Paris) or Foch Hospital (Suresnes).

* Close relatives of lung transplant patients (spouse; partner; first-degree parent) followed at Bichat Hospital (Paris) or Foch Hospital (Suresnes).
* Physicians from lung transplant centers in France, or French-speaking experts identified in the professional network of investigators.
* Paramedical staff (state certified nurses, psychologists, physiotherapists, etc.) from the same French center or French-speaking centers whose primary focus is on caring for lung transplant patients.

Exclusion Criteria:

* Patients or close relatives under guardianship or protective supervision.
* Minor patients or minor close relatives.
* Patients or close relatives of recently transplanted patients (immediate post-transplant hospitalization).
* Patients or close relatives of patients who have undergone a combined transplant (liver-lung, heart-lung, kidney-lung).
* Non-comprehension of the French language.
* Inability to use computer tools.
* Refusal to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Lung transplant patients
  * Relatives of lung transplant patients
  * Physicians
  * Pramedical staff
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Identifying a set of outcome criteria defined as Patient Important Outcomes (PIO) from the perspective of physicians, paramedics, lung transplant patients, and their families | 3 weeks
  Delphi method

SECONDARY OUTCOMES:
Evaluate the participation within each panel and at each round of the Delphi survey. | 3 weeks
  Rate of participation within each panel and at each round of the Delphi survey.

CONTACTS AND LOCATIONS:
Overall Officials: WEISENBURGER Gaëlle, MD, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX DE PARIS-Hôpital Bichat